CLINICAL TRIAL: NCT06886906
Title: Exploring the Acute and Dynamic Relationships Between Movement and Pain in Older Adults With Musculoskeletal Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kelly Naugle, PhD, Associate Professor, Indiana University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 24426
Record Dates: First submitted 2025-03-14; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Older People; Pain
Keywords: physical activity; movement evoked pain; sitting; quantitative sensory testing; musculoskeletal pain
MeSH Terms: conditions — Pain; Motor Activity; Musculoskeletal Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uninterrupted Sitting for 1 hour (Experimental): The participant will remain seated throughout the experimental period and will be instructed to minimize excessive movement, only rising from the chair to void. This experimental condition is designed to mimic prolonged uninterrupted sedentary behavior.
  Interventions: Behavioral: uninterrupted sitting
- 1 hour of sitting interrupted with 2.5 minute bouts of light intensity walking (Experimental): Participants will sit as described above with six bouts of 2.5-minutes of light intensity walking (see Figure 2). Overall, the bouts will occur on six occasions, providing a total of 15 minutes of light intensity activity. Participants will be asked to walk at a light intensity based on the 6-20 RPE scale, which corresponds to a 9-11 RPE rating. This experimental condition is designed to mimic sedentary behavior interspersed with frequent short bouts of LPA. RPE and pain intensity (0-100 scale) will be assessed at the end of each walking bout.
  Interventions: Behavioral: Intermittent light walking

INTERVENTIONS:
Behavioral: Intermittent light walking — The participant will remain seated throughout the 1 hour experimental period. During this 1-hour period, participants will complete six bouts of 2.5-minutes of light intensity walking. Overall, the bouts will occur on six occasions, providing a total of 15 minutes of light intensity activity.
  Other Names: 1 hour of sitting interrupted with 2.5 minute bouts of light intensity walking
  Arms: 1 hour of sitting interrupted with 2.5 minute bouts of light intensity walking
Behavioral: uninterrupted sitting — The participant will remain seated throughout the experimental period and will be instructed to minimize excessive movement, only rising from the chair to void. This experimental condition is designed to mimic prolonged uninterrupted sedentary behavior.
  Arms: Uninterrupted Sitting for 1 hour

SUMMARY:
The purpose of this research study is to evaluate the effect of brief bouts of intermittent walking on bodily pain, pain during movement, and how the body adapts to musculoskeletal pain in older adults.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether exposure to acute sitting compared to sitting interrupted with brief bouts of light intensity walking exerts short term effects on resting pain, endogenous pain modulation measured via quantitative sensory testing (QST), and movement-evoked pain (MEP) in older adults. Participants will be asked to complete two study sessions, with the first study session lasting 3 hours and the second study session lasting 2.5 hours. All sessions will take place in the National Institute of Sport Fitness, where the Physical Activity and Pain laboratory is located. The first session will include the following procedures in the following order: informed consent process, healthy history for screening purposes, quantitative sensory testing (QST), 6-minute walk test, completion of questionnaires, QST, experimental conditions of either 1 hour of sitting or 1 hour of sitting with bouts of light intensity walking, QST, and the 30-second chair stand test. Session 2 will take place at least 7 days after session 1 and will be identical except for the informed consent and screening will be replaced by questionnaires and the experimental condition will consist of the one not performed in session 1. Participants will be asked to take their medications at the same time prior to each study visit and we will assess medications taken the day of each visit prior to the visit.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling men and women
* Answer yes to the following question: Have you experienced any musculoskeletal pain (pain affecting joints, bones, ligaments, tendons or muscles) in the past month?

Exclusion Criteria:

* Cardiovascular issues such as uncontrolled blood pressure over 150/99 mmHg, heart failure, or history of acute myocardial infarction;
* Angina in the last month (squeezing, pressure, heaviness, tightness, or pain in chest)
* Serious systemic disease or condition (e.g., severe osteoarthritis, injury) that restricts normal daily activities
* Neurological disease (e.g., Parkinson's Disease, multiple sclerosis, epilepsy)
* Serious psychiatric conditions (schizophrenia, bipolar disorder) or hospitalization within the preceding year for psychiatric illness
* Known peripheral neuropathy
* Chronic opioid use (defined as ≥ 90 days)
* Unable to walk for 6 minutes without assistive devices

Session exclusion criteria:

• Participants will be asked to not participate in vigorous or unaccustomed exercise 48 hours prior to each study session.

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Mechanical Temporal Summation of Pain (TS) | Pre and post the 1-hour experimental conditions
  TS will be administered on the back of the left hand. First, a single pinprick stimulus using a von Frey filament of 6.65 Mn or 300 g will be applied to the body site. Participants will rate the perceived pain intensity using a numeric rating scale of 0 (no pain at all) to 100 (worst pain imaginable). Then, a series of 10 pinprick stimuli (6.65 Mn) will be administered at a rate of 1 Hz, applied to the body site within an area of 1 cm2. The temporal summation value will be calculated as the difference between the first and last stimuli.
Conditioned Pain Modulation | Pre and post the 1-hour experimental conditions
  CPM will be assessed by determining the ability of a cold water bath (conditioning stimulus) to diminish pressure pain thresholds (PPTs) and temporal summation (TS) (test stimuli) applied at a separate body site. For the CPM trials, PPTs and TS will be measured pre and post a conditioning stimulus. Conditioning stimulus: At least 4 minutes will separate the pre pain assessments (i.e., PPT, TS) and the initiation of the conditioning stimulation, during which subjects will sit quietly. Then, participants will immerse their right hand up to the wrist in a cold water bath maintained at 10oC for up to 1 minute or until they report intolerable pain. The dependent variable for the CPM test will be the change in the test stimuli (PPT and TS) following the conditioning stimulus.
Movement-evoked pain during the 30-second chair stand test | Will be administered immediately after the 1-hour experimental conditions.
  This test will be administered using a folding chair without arms, placed against a wall to prevent it from moving during the test. The test begins with the subject seated in the middle of the chair, feet at an angle slightly back from the knees, with one foot slightly in front of the other to help maintain balance when standing. Arms will be crossed at the wrists and held against the chest. At the signal of "go", subjects will rise to a full stand and then return back to the initial position. The subjects will be encouraged to complete as many full stands as possible within a 30-s time limit. Participants will rate their current bodily pain on a 0 to 10 numeric rating scale (NRS), with 0 indicating "No pain" and 10 indicating "Pain as bad as you can imagine". Participants will rate their bodily pain before, during, and after the chair stand test as a measure of movement evoked pain.

OTHER OUTCOMES:
Physical Activity and Sedentary Behavior Questionnaire (PASB-Q) | At baseline during one of the study sessions
  The PASB-Q has 7 items to measure reported aerobic PA, muscle strengthening PA, perceived aerobic fitness, and sedentary behavior.
The Physical Activity Scale for the Elderly (PASE) | At baseline during one of the study sessions
  The PASE has a total of 18 items using a 4-point scales and yes/no questions. The items capture seven dimensions of physical activity. People with higher scores are more physically active.
Movement evoked pain during the six minute walk test | At baseline during each study session.
  Subjects will be required to walk as far as possible at their usual pace in 6 minutes around a predetermined indoor walking course on a flat surface. The distance subjects cover will be recorded. Participants will rate their current bodily pain on a 0 to 10 numeric rating scale (NRS), with 0 indicating "No pain" and 10 indicating "Pain as bad as you can imagine". Participants will rate their bodily pain before, during, and after the walk as a measure of movement evoked pain.
Graded Chronic Pain Scale (GCPS) | At baseline during one of the study sessions
  The GCPS will be used to measure pain-related severity and disability across 7-items
Pain Catastrophizing Scale (PCS) | At baseline during one of the study sessions
  The PCS asks the respondents to reflect upon past painful experiences and to rate the degree to which they experienced negative thoughts or feelings about pain. Catastrophizing is a multidimensional construct composed of rumination, helplessness, and magnification.
Short-Form Health Survey-36 (SF-36) | At baseline during one of the study sessions
  The SF-36 is a health survey that yields 8-scale scores (physical functioning, role limitations due to physical problems, bodily pain, vitality, general health perceptions, social functioning, role limitations due to emotional problems, and mental health).
Tampa Scale of Kinesiophobia (TSK) | At baseline during one of the study sessions
  The TSK consists of 11 items and is rated on a 4-point scale. The TSK is used to measure the fear of movement or re-injury. The TSK has been deemed a valid and reliable method for determining fear of movement in both clinical and nonclinical populations.
Pain Disability Index (PDI) | At baseline during one of the study sessions
  The PDI is a simple and rapid 7-item instrument for measuring the impact that pain has on the ability of a person to participate in essential life activities.
Anatomical map for locating pain areas | At baseline during one of the study sessions
  We will use an anatomical map for locating pain areas that is part of the Pain Assessment Screening Tool and Outcomes Registry (PASTOR).
Pittsburgh Sleep Quality Index (PSQI) | At baseline during one of the study sessions
  The PSQI is a self-report questionnaire used to assess sleep quality and quantity over the last month. The PSQI includes 19 items to measure seven domains of sleep quality: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, daytime dysfunction, sleep disturbance and use of sleeping medications.
Adult Hope Scale (AHS) | At baseline during one of the study sessions
  AHS is a measure of trait hope in adults formed from agency and pathways thinking. The AHS includes 12 statements that participants rate from 1 (definitely false) to 8 (definitely true) for how the statements describe them. (e.g., "I can think of many ways in life to get the things that are most important to me").
Ratings of perceived exertion (RPE) | During the intermittent bouts of walking during the walking experimental condition
  Subjects will rate their perception of exertion while walking using Borg's RPE scale. This rating should reflect how heavy and strenuous the exercise feels, combining all sensations and feeling of physical stress, effort, and fatigue. The scale ranges from 6 to 20, where 6 means "no exertion at all" and 20 means "maximal exertion."

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Marie Naugle, Principal Investigator — School of Health and Human Sciences, IUPUI
Locations (1):
- 250 University Blvd, Indianapolis, Indiana, United States